CLINICAL TRIAL: NCT03390517
Title: A Study of Perfusion of Colorectal Anastomosis Using FLuorescence AnGiography (FLAG-trial)
Acronym: FLAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State Scientific Centre of Coloproctology, Russian Federation (Other Government)
Responsible Party: Principal Investigator, Rybakov Evgeny, MD, Dr.Med.Sc. State Scientific Centre of Coloproctology, Head of Surgical department of oncoproctology, Moscow, Russian Federation, State Scientific Centre of Coloproctology, Russian Federation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 80
Record Dates: First submitted 2017-12-27; First posted 2018-01-04 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Rectal Cancer; Sigmoid Cancer
Keywords: fluorescence angiography; indocyanine green; anastomotic leakage
MeSH Terms: conditions — Rectal Neoplasms; Sigmoid Neoplasms; Anastomotic Leak | interventions — Fluorescein Angiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICG group (Experimental): A sigmoid and rectum resection with colorectal anastomosis will be performed according to the surgeons standard practice with the addition of intraoperative imaging using fluorescence angiography with indocianyne green to assess colon and rectal tissue perfusion.
  Interventions: Device: Fluorescence angiography with indocianyne green
- Standard (No Intervention): A sigmoid and rectum resection with colorectal anastomosis will be performed according to the surgeons standard practice.

INTERVENTIONS:
Device: Fluorescence angiography with indocianyne green — The fluorescence angiography was performed after mobilization of the bowel, transection of the rectum, division of the rectal and colon mesentery and central vessels, before specimen extraction or resection and creation of the anastomosis. This site was selected by the surgeon using his or her best judgment and typical standard of care assessment. After this selection, the anesthesiologist administered a bolus of 1 to 2 ml indocianyne green intravenously. Perfusion of the colon was visualized and assessed via fluorescence angiography and the line of demarcation between perfused and nonperfused tissue was noted and compared with the initial planned transection point.
  Arms: ICG group

SUMMARY:
This is a randomized, controlled, parallel study to determine the difference in post-operative anastomotic leak rate of colorectal anastomosis where colon and rectal tissue perfusion is evaluated using fluorescence angiography with indocyanine green and without this method.

DETAILED DESCRIPTION:
The design involves random allocation of eligible patients to operation with colorectal anastomosis and intraoperative fluorescence angiography with indocyanine green and operation alone. After surgery on 7-8 POD patients are examined to two sides X-Ray proctography performed by introducing 100 ml of water-soluble liquid contrast material through the anus over the anastomotic line by a Foley catheter for diagnosis of anastomotic leakage.

ELIGIBILITY:
Inclusion Criteria:

* Have a planned circular stapled colorectal anastomosis
* Have signed an approved informed consent form for the study

Exclusion Criteria:

* Has known allergy or history of adverse reaction to indocianyne green, iodine or iodine dyes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 18 years and older
Enrollment: 377 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2019-09-22 (Actual)

PRIMARY OUTCOMES:
Anastomotic Leak Rate | 0 to 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- State Scientific Centre of Coloproctology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No